CLINICAL TRIAL: NCT03369457
Title: Analysis of the Osteogenic Potential of Multipotent Cells From Different Anatomical Regions in Hip Replacement Surgery
Brief Title: Analysis of the Osteogenic Potential of Multipotent Cells From Different Anatomical Regions
Acronym: EMPHA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: EMPHA
Record Dates: First submitted 2017-12-06; First posted 2017-12-12 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Complications; Implant, Orthopedic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Mesenchymal stromal cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Isolation of multipotent cells — Isolation of multipotent cells from patient's cells. Analysis of CFU and differentiation potential

SUMMARY:
The aim of hip replacement surgery is to re-establish the physiological hip function and to obtain a stable fixation between the prosthetic components and the native bone. Commonly, the fixation is obtained by bone ingrowth between the prosthesis and the native bone. Thus, the quality of the patient's bone stock is essential to achieve this aim. However, several clinical conditions may impair the bone stock; therefore, in these cases bone grafts are necessary to improve the prosthetic fixation. The gold standard is represented by autologous bone grafts (from iliac crest or from acetabular bone chips) or allogeneic bone grafts from cadaveric femoral heads. Nevertheless, the osteogenic potential of multipotent cells derived from different anatomical regions has never been examined.

Thus, the aim of this study is to isolate multipotent cells from acetabular or femoral bone chips and from bone marrow aspirate of the same patient and to compare their osteogenic potential. The results of this study may reveal differences, which may have a clinical relevance for hip replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hip replacement and affected by:

  1. hip osteoarthritis
  2. mild developmental dysplasia of the hip
* 18 ≤ Body Mass Index (BMI) ≤ 30 kg/m2

Exclusion Criteria:

* Rheumatoid arthritis
* Patients under pharmacological treatment for bone metabolic disorders
* Patient affected by metabolic disorders, which may affect bone metabolism
* Presence of bone metastases
* Presence of bone infections
* Patients undergoing hip revision surgeries
* Obesity (BMI ≥30kg/m2)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 13 patients undergoing hip replacement surgery will be selected. Samples from acetabulum, proximal femur (head of the femur) and from bone marrow will be collected for each patient.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Estimated)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2020-06-14 (Estimated)

PRIMARY OUTCOMES:
Evaluation of differences in Colony Forming Units (CFU) percentage | 6 months
  Formation of CFUs will be evaluated in the three different samples (acetabular bone chips, femoral bone chis or bone marrow aspirated) and CFUs will be counted in each sample

SECONDARY OUTCOMES:
Evaluation of the osteogenic potential in the three different cell populations | 1 year
  Evaluation of Alizarin red stain. Analysis of bone markers (RUNX2, Collagen type I, Collagen type X, Alkaline Phosphatase)
Evaluation of the chondrogenic potential in the three different cell populations | 1 year
  Evaluation of Alcian blue stain in pellet culture. Analysis of chondrogenic markers (Collagen type II and SOX9)
Evaluation of the adipogenic potential in the three different cell populations | 1 year
  Evaluation of Oil red stain. Analysis of adipogenic markers (Peroxisome proliferator-activated receptor gamma (PPAR-γ), Lipoprotein lipase (LPL))

CONTACTS AND LOCATIONS:
Overall Officials: Laura Mangiavini, Principal Investigator — IRCCS Istituto Ortopedico Galeazzi
Locations (1):
- IRCCS Istituto Ortopedico Galeazz, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen VT, Tessaro I, Marmotti A, Sirtori C, Peretti GM, Mangiavini L. Does the Harvesting Site Influence the Osteogenic Potential of Mesenchymal Stem Cells? Stem Cells Int. 2019 May 2;2019:9178436. doi: 10.1155/2019/9178436. eCollection 2019. PMID 31191688